CLINICAL TRIAL: NCT07160140
Title: Investigation of the Effect of Pedal Technique Training Protocol on Functional Threshold Power Test and Lower Extremity Isokinetic Power
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Topkapi University (Other)
Responsible Party: Principal Investigator, Aliye Buyukergunkaplan, Assistant Professor, Istanbul Topkapi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: E-74555795-050.01.04-392011
Record Dates: First submitted 2025-08-24; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Isokinetic Test; Cyclists; Performance Enhancement
Keywords: Pedal technique, Bicycle, Isokinetic power, Assymetry, Functional threshold power

STUDY DESIGN:
Intervention Model Description: In this study, a fully experimental research method was followed using a pre-test-post-test research design with a predetermined control group. The experimental method refers to a type of research that includes the processes of applying the factor to be examined to the participants under certain rules and conditions, measuring the reactions of the participants to the factor, and reaching conclusions by comparing the assembled results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group - Pedal Technique Training (Active Comparator): Participants will receive an 8-week pedal technique training protocol in addition to their regular cycling training.
  Interventions: Other: Participants will receive an 8-week pedal technique training protocol in addition to their regular cycling training.
- Control - Usual Training (No Intervention): Participants will continue their regular cycling training without any additional intervention.

INTERVENTIONS:
Other: Participants will receive an 8-week pedal technique training protocol in addition to their regular cycling training. — Pedal Technique Training Protocol This training is designed as a technical training to observe pedaling data, analyze right and left leg power ratios, and determine how they change when pedaling at various intensities and cadences
  Arms: experimental group - Pedal Technique Training

SUMMARY:
Abstract Purpose: The objective of this study is to assess the influence of pedal technique development training regimen on functional threshold power, lower extremity knee isokinetic power, and right-left knee power ratio differences.

Methods: Twenty-three male athletes with an average age of 15-17 years in the youth division of road cycling voluntarily participated in the study. Within the scope of the study, height, body weight, body fat ratio measurements, functional threshold power, pedal analysis tests, and lower extremity knee power measurements were performed as pre-test and post-test. Athletes participated in an 8-week, two-day-per-week pedal technique development training program. Statistical analyses were planned to be carried out on the data gathered from these measurements, calculations, and tests.

DETAILED DESCRIPTION:
The study included 24 male athletes between the ages of 15-17 who continue their sports careers at the national team level. The participants consisted of a total of 24 athletes, 12 in the training group and 12 in the control group.

The research program was carried out two days a week for 8 weeks. During this period, the experimental group received their own bicycle training programs in addition to pedal technique development training, while the control group continued their regular bicycle training only. The study was designed as an experimental research with a pre-test-post-test design and a predetermined control group. The experimental approach refers to applying the factor to be investigated under specific rules and conditions, evaluating the participants' responses, and then analyzing the data obtained.

The study was divided into three phases: pre-testing, training, and post-testing. It lasted eight weeks. During the pre-test and post-test periods, both the training and control groups underwent one week of assessments.

The ethical suitability of the study within the scope of scientific research was examined by the Presidency of the IUC Non-Interventional Clinical Research Ethics Committee, and approval was obtained with the decision letter dated 22.05.2022 and numbered E-74555795-05.01.04-392011.

ELIGIBILITY:
Inclusion Criteria:

* Male youth athletes aged 15-17 years
* Registered in a road cycling team
* Minimum 2 years of continuous cycling training experience
* Voluntary participation and informed consent

Exclusion Criteria:

* Musculoskeletal injury in the past 6 months
* Chronic diseases affecting performance
* Participation in another intervention study within the past 3 months

Ages: 15 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — male
Enrollment: 24 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Functional Threshold Power (W/kg) as Measured by Standardized Cycling Test | Baseline and 8 weeks
  Functional Threshold Power (FTP) will be assessed using a standardized cycling protocol on a road bike trainer. The change from baseline to post-intervention (8 weeks) will be analyzed.

SECONDARY OUTCOMES:
Change from Baseline in Knee Extension Peak Torque at 60°/sec | Baseline and 8 weeks
  Knee extension peak torque will be measured at an angular velocity of 60°/sec using an isokinetic dynamometer. Changes from baseline to 8 weeks will be analyzed.
Change from Baseline in Knee Flexion Peak Torque at 60°/sec | Baseline and 8 weeks
  Knee flexion peak torque will be measured at an angular velocity of 60°/sec using an isokinetic dynamometer. Changes from baseline to 8 weeks will be analyzed.
Change from Baseline in Knee Extension Peak Torque at 180°/sec | Baseline and 8 weeks
  Knee extension peak torque will be measured at an angular velocity of 180°/sec using an isokinetic dynamometer. Changes from baseline to 8 weeks will be analyzed.
Change from Baseline in Knee Flexion Peak Torque at 180°/sec | Baseline and 8 weeks
  Knee flexion peak torque will be measured at an angular velocity of 180°/sec using an isokinetic dynamometer. Changes from baseline to 8 weeks will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Topkapi University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including baseline characteristics, intervention details, and outcome measures) will be shared for research purposes upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The dataset will be available beginning 6 months after publication and ending 5 years after study completion.
Access Criteria: Researchers who provide a methodologically sound proposal and obtain ethical approval may access the data through a secure data repository.